CLINICAL TRIAL: NCT01480479
Title: An International, Randomized, Double-Blind, Controlled Study of Rindopepimut/GM-CSF With Adjuvant Temozolomide in Patients With Newly Diagnosed, Surgically Resected, EGFRvIII-positive Glioblastoma
Brief Title: Phase III Study of Rindopepimut/GM-CSF in Patients With Newly Diagnosed Glioblastoma
Acronym: ACT IV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDX110-04
Record Dates: First submitted 2011-11-21; First posted 2011-11-29 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2017-04

CONDITIONS: Glioblastoma; Small Cell Glioblastoma; Giant Cell Glioblastoma; Gliosarcoma; Glioblastoma With Oligodendroglial Component
Keywords: EGFRvIII; Glioblastoma; Small cell; Giant cell; Gliosarcoma; oligodendroglial; Brain Cancer; Brain Tumor; radiotherapy; chemoradiation; Tumor; temozolomide; EGFR variant III
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms; Neoplasms | interventions — rindopepimut; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Temozolomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rindopepimut/GM-CSF plus Temozolomide (Experimental)
  Interventions: Drug: Rindopepimut (CDX-110) with GM-CSF; Drug: Temozolomide
- KLH plus Temozolomide (Active Comparator)
  Interventions: Drug: Temozolomide; Drug: KLH

INTERVENTIONS:
Drug: Rindopepimut (CDX-110) with GM-CSF — Two intradermal injections two weeks apart, followed by monthly injections until tumor progression or intolerance.
  Each dose will be 0.8 mL containing approximately 500 mcg CDX-110 and 150 mcg GM CSF.
  Other Names: CDX-110 with sargramostim (GM-CSF) (Leukine®)
  Arms: Rindopepimut/GM-CSF plus Temozolomide
Drug: Temozolomide — 150 to 200 mg/m2 for 5 days during each 28-day cycle for a minimum of six cycles or a maximum of 12 cycles, or until intolerance or progression.
  Other Names: Temodar; Temodal
Drug: KLH — Two intradermal injections two weeks apart, followed by monthly injections until tumor progression or intolerance. Each dose will be 0.8mL containing approximately 100mcg of KLH.
  Arms: KLH plus Temozolomide

SUMMARY:
This 2-arm, randomized, phase III study will investigate the efficacy and safety of the addition of rindopepimut (an experimental cancer vaccine that may act to promote anti-cancer effects in patients who have tumors that express the EGFRvIII protein) to the current standard of care (temozolomide) in patients with recently diagnosed glioblastoma, a type of brain cancer.

All patients will be administered temozolomide, the standard treatment for glioblastoma. Half the patients will be randomly assigned to receive rindopepimut and half the patients will be randomly assigned to receive a control called keyhole limpet hemocyanin.

Patients will be treated in a blinded fashion (neither the patient or the doctor will know which arm of the study the patient is on). Patients will be treated until disease progression or intolerance to therapy and all patients will be followed for survival.

DETAILED DESCRIPTION:
The purpose of this research study is to find out whether adding an experimental vaccine called rindopepimut (also known as CDX-110) to the commonly used chemotherapy drug temozolomide can help improve the life expectancy of patients with newly diagnosed, resected EGFRvIII positive glioblastoma.

The duration of participation in this study may be up to 5 years. After you are screened and enrolled in the study, you will be administered temozolomide and either rindopepimut/GM-CSF or KLH until either disease progression or intolerance to the medications. If your tumor progresses while on this study, your doctor may treat you with other therapies that are not part of the study.

ELIGIBILITY:
Inclusion Criteria-

Among other criteria, patients must meet the following conditions to be eligible for the study:

1. Adult patients, ≥ 18 years old
2. Newly diagnosed glioblastoma
3. Attempted surgical resection followed by conventional chemoradiation
4. Documented EGFRvIII positive tumor status by a Sponsor designated laboratory
5. No evidence of progressive disease from the post-operative period to the post-chemoradiation period
6. Candidate for, and agrees to receive, adjuvant (maintenance) temozolomide therapy
7. Systemic corticosteroid therapy at ≤2 mg of dexamethasone or equivalent per day for at least 3 days prior to randomization
8. WHO-ECOG Performance Status ≤ 2
9. Patients of childbearing/reproductive potential will be instructed to use birth control as defined by your doctor.

Exclusion Criteria-

Among other criteria, patients who meet the following conditions are NOT eligible for the study:

1. Stereotactic biopsy only (without further surgical resection)
2. Presence of diffuse leptomeningeal disease, gliomatosis cerebri, or infratentorial disease.
3. History, presence, or suspicion of metastatic disease
4. Patients who have received any additional treatment for glioblastoma, aside from surgical resection and chemoradiation with temozolomide
5. Active systemic infection requiring treatment
6. History of any malignancy (other than glioblastoma) during the last three years except non-melanoma skin cancer, in situ cervical cancer, treated superficial bladder cancer, cured, early-stage prostate cancer in a patient with PSA level less than ULN,or other carcinoma in situ that has been adequately treated and cured.
7. Planned major surgery
8. Evidence of current drug or alcohol abuse
9. Known allergy or hypersensitivity to keyhole limpet hemocyanin (KLH), GM-CSF (sargramostim; LEUKINE®), polysorbate 80 or yeast derived products, or a history of anaphylactic reactions to shellfish proteins
10. Severe acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with participating in a clinical trial
11. Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 745 (Actual)
Dates: Start 2011-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Overall Survival | During treatment and every three months from end of treatment through end of study or approximately up to 5 years.
  The primary efficacy endpoint of Overall Survival is defined as the number of months from randomization to the date of death (whatever the cause), and will be censored for patients who remain alive at completion of the study for patients with a gross total resection (~n=374). The overall survival of patients will be monitored and compared between the two study arms until the end of the study.

SECONDARY OUTCOMES:
Progression-free survival | Every 12 weeks from Day 1 through progression or initiation of other anti-cancer therapy
  Compare progression-free survival between the two treatment arms
Safety and Tolerability | Until day 28 of follow up
  Safety and tolerability will be measured by comparing the two arms in regards to vital sign measurement, physical and neurological examination, adverse events reporting, ECOG performance status, and EORTC core Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Locations (223):
- United States (88):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Barrow Neurological Institute at St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of Arizona Health Network, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente, Redwood City Medical Center, Redwood City, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Stanford Cancer Institute, Stanford University, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale University Medical Center, New Haven, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - University of Florida, Gainesville, Florida
  - Mount Sinai Medical Center, Comprehensive Cancer Center, Miami Beach, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Atlanta Cancer Care, Atlanta, Georgia
  - Winship Cancer Institute, Emory University School of Medicine, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Kaiser Permanente Hawaii Moanalua Medical Center, Honolulu, Hawaii
  - Northwestern University Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - North Shore University Health System, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Covenant Clinic / Iowa Spine and Brain Institute, Waterloo, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - LSU Health Sciences Center, Feist-Weiller Cancer Center, Shreveport, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, PC, Bethesda, Maryland
  - Dana-Farber Cancer Institute and Mass General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Edward W. Sparrow Hospital Association - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary's of Michigan Medical Center/Field Neurosciences Institute, Saginaw, Michigan
  - Allina Health, Abbott Northwestern Hospital, John Nasseff Neuroscience Institute, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - New Jersey Neuroscience Institute, JFK Medical Center, Edison, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Dent Neurosciences Research Institute, Amherst, New York
  - New York Methodist Hospital, Brooklyn, New York
  - The Long Island Brain Tumor Center at Neurology Surgery, P.C., Great Neck, New York
  - North Shore University Hospital, Manhasset, New York
  - Columbia University Medical Center - The Neurologic Institute of New York, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Brain and Spine Surgeons of New York, White Plains, New York
  - The Preston Robert Tisch Brain Tumor Center at Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - University Hospitals, Case Medical Center (Cleveland), Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Providence Portland Medical Center, Oncology & Hematology Care, Portland, Oregon
  - Pacific Neurosurgical, Portland, Oregon
  - Lehigh Valley Physician Group-Hematology-Oncology Associates, Allentown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - West Penn. Allegheny Health System, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Medical University of South Carolina - Department of Neuroscience, Charleston, South Carolina
  - University of Tennessee Medical Center - Knoxville, Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology Midtwon, Austin, Texas
  - Baylor Research Institute, Dallas, Texas
  - The Methodist Neurological Institute, Houston, Texas
  - University of Utah Department of Neurosurgery, Salt Lake City, Utah
  - Fletcher Allen Health Care, Burlington, Vermont
  - University of Virginia Healthcare System, Charlottesville, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Paul P Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (14):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Crown Princess Mary Cancer Centre, Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Adult Hospital, Mater Misericordiae Health Services Brisbane Limited, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Calvary North Adelaide Hospital, North Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital, Launceston, Tasmania
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Epworth Healthcare, Richmond, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Liverpool Hospital, Liverpool
- Austria (2):
  - Medical University Innsbruck, Dept of Neurology, Anichstrabe 35, Innsbruck
  - Medizinische Universität Wien, Innere Medizin I, Onkologie, Vienna
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerp
  - ZNA Middelheim, Antwerp
  - Ghent University Hospital, Ghent
- Brazil (8):
  - Hospital Mae de Deus-Centro de Pesquisa em Oncologia Clinica, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Clinicas da Fundação Dr Amaral Carvalho, Jaú, São Paulo
  - Fundação Faculdade Regional de Medicina de de São José do Rio Preto - Hospital de Base, São José do Rio Preto, São Paulo
  - Instituto Nacional do Cancer (INCA), Rio de Janeiro
  - Instituto do Câncer do Estado de São Paulo - ICESP, São Paulo
  - Real e Benemerita Associação Portuguesa de Beneficiência/ Hospital São José, São Paulo
  - Hospital A C Camargo, São Paulo
  - Hospital Albert Einstein, São Paulo
- Canada (13):
  - Foothills Hospital Medical Centre, Calgary, Alberta
  - British Columbia Cancer Agency, Vancouver Clinic, Vancouver, British Columbia
  - BC Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - University of Manitoba-Cancer Care Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program, London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Regional Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM) - Hopital Notre-Dame, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - CHUQ L'Hotel Dieu de Qujebec, Québec, Quebec
  - CHUS Hôpital Fleurimont, Shenbrooke, Quebec
- Fundacion Santa Fe, Bogotá, Bogota D.C., Colombia
- Czechia (5):
  - Hospital Ceske Budejovice, České Budějovice
  - Umiversity Hospital (Fakultni Nemocnice), Prague
  - Hospital Na Homolce, Prague
  - Multiscan s.r.o., Prague
  - Masaryk´s Hospital Usti nad Labem, Ústí nad Labem
- France (9):
  - Institut de Cancerologie de I'Quest-Paul Papin, Angers
  - Institute Bergonie, Bordeaux
  - Centre Leon Berard de Lyon, Lyon
  - ICM Val d'Aurel Montpellier, Montpellier
  - Institut de Cancerologie de L'Quest-Center Rane Gauducheau, Nantes
  - Service de Neurologie-GH, Paris
  - Centre Eugene Marquis, Rennes
  - Institut de Cancerologie de l'ouest-Center Rene Gauducheau, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Germany (8):
  - Klinik und Poliklinik fur Neurologie der Universitat Regensburg, Regensburg, Bavaria
  - Strahlenklinik Universitatsklinikum Erlangen, Erlangen
  - Dr. Senchkenbergisches Institut fur Neuroonkologie, Frankfurt
  - University Hospital Hamburg Kopf und Neurozentrum, Hamburg
  - Universitaetsklinikum Heidelberg, Neurologische Klinik, IM Neuenheimer Feld 672, Heidelberg
  - University Medical Centre, Kiel
  - LMU Munich, Munich
  - Universitaetsklinikum Muenster, Münster
- Greece (2):
  - NNA, Athens, Attica
  - "HYGEIA" Hospital, Marousi, District of Attica
- Hungary (6):
  - Országos Onkológiai Intézet Sugárterápiás Osztály, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum Onkológiai Intézet, Debrecen
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Sugárterápiás Osztály, Miskolc
  - Pécsi Tudományegyetem Általános Orvostudományi Kar, Pécs
  - Szegedi Tudományegyetem Onkoterápiás Klinika, Szeged
  - Vas Megyei Markusovszky Lajos Általános Rehabilitációs és Gyógyfürdő Kórház, Egyetemi Oktatókórház Nonprofit Zrt, Szombathely
- India (11):
  - City Cancer Centre, Vijayawada, Vijayawada, Andhra Pradesh
  - HCG - Bangalore Institute of Oncology, Bangalore, Bengaluru, Karnataka
  - Amrita Institute of Medical Sciences and Research Centre, Kochi, Kochi, Kerala
  - Sree Chitra Tirunal Institute for Medical Sciences & Technology, Thiruvananthapuram, Thiruvananthapuram, Kerala
  - Marathwada Regional Cancer Centre and Research Institute - Government, Aurangabad, Maharashtra
  - Kokilaben Dhirubhai Ambani Hospital and Medical Research Institute, Andheri-West, Mumbai
  - Tata Memorial Hospital , Mumbai, Pārel, Mumbai
  - Indraprastha Apollo Hospital, New Delhi, Jasola Viha, New Delhi
  - Sahyadri Hospitals Limited, Erandauame, Pune
  - Dr. Rai Memorial Medical Centre, Chennai, Chennai, Tamil Nadu
  - HCG Shanti Mukand Hospital - Curie Cancer Centre, Delhi, Delhi
- Israel (5):
  - Soroka University M.C., Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - SHEBA Medical Center, Tel Litwinsky
- Italy (4):
  - UO Oncologie Medica Dipartimento Oncologico, Bologna
  - Fondazione IRCCS Instituto Neurologico Carlo Besta, Milan
  - Sacred Heart Catholic University, Rome
  - Universita e AO Citta delia Scienza, Universita Di Torino, Torino
- Mexico (5):
  - Grupo Médico Camino S.C., México, D.F
  - Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco
  - Ensayos Clínicos y Medicina de Alta Especialidad, S.C., Culiacán, Sinaloa
  - Servicios Medicos de Investigacion Clinica Sc, Durango
  - Hospital Central "Ignacio Morones Prieto", San Luis Potosí City
- Netherlands (3):
  - Medisch Centrum Haaglanden, The Hague, South Holland
  - VUMC, Amsterdam
  - Radboud University Nijmegen Medical Center, Nijmegen
- New Zealand (4):
  - Christchurch Hospital, Christchurch Central, Christchurch
  - Palmerston North Hospital, Roslyn, Palmerston North
  - Waikato Hospital, Regional Cancer Centre, Hamilton, Waikato District
  - Waikato Hospital, Regional Cancer Center, Hamilton, Waikato Distric
- Peru (5):
  - Hospital Almanzor Aguinaga Asenjo, Chiclayo
  - Instituto Oncologico Miraflores, Lima
  - Clinica Anglo Americana, Lima
  - Clinica Ricardo Palma, Lima
  - Oncosalud, Lima
- Spain (5):
  - Institut Catala d Oncologia, LaHospitalet de Lubregat, Catalonia
  - Dra. Sonia Del Barco Berron, ICO Girona Avda,, Franca, Girona
  - Hospital Clinic, Barcelona
  - ICO Badalona-Hospital Germans Trias i Pujol, Barcelonia
  - Hospital 12 de Octubre, Madrid
- Switzerland (6):
  - Kantonsspital Aarau Medizinische Onkologie Tellstrasse, Aarau, Canton of Aargau
  - CHUV, Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - Oncology Institute of Southern Switzerland (IOSI), Bellinzona
  - Inselspital, Universitatsspital Bern, Universitatsklinik fur Medizinische Onkologie, Freiburgstrasse, Bern
  - Hopitaux Universitaires de Geneve-HUG-Centre d'Oncologie, Geneva
  - Brain Tumor Center, University Hospital Zurich, Zurich
- Taiwan (6):
  - National Cheng Kung University Hospital, Tainan, Bei District
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Linkou Branch, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Tainan City - Yongkang District
  - Tri-Service General Hospital, Taipei City - Neihu District
- Thailand (4):
  - Siriraj Hospital, Bangkoknoi, Bangkok
  - King Chulalongkorn Memorial Hospital, Patumwan, Bankok
  - Songkhlanagarind Hospital, Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital, Amphoe Muang, Chiang Mai
- United Kingdom (6):
  - Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - The Bristol Haematology and Oncology Centre, Bristol
  - Edinburgh Cancer Centre Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centrel, Glasgow
  - Guy's and St Thomas' NHS, Westminister Bridge Road, London
  - Nottingham City Hospital, Nottingham

REFERENCES:
- [Result] Weller M, Butowski N, Tran DD, Recht LD, Lim M, Hirte H, Ashby L, Mechtler L, Goldlust SA, Iwamoto F, Drappatz J, O'Rourke DM, Wong M, Hamilton MG, Finocchiaro G, Perry J, Wick W, Green J, He Y, Turner CD, Yellin MJ, Keler T, Davis TA, Stupp R, Sampson JH; ACT IV trial investigators. Rindopepimut with temozolomide for patients with newly diagnosed, EGFRvIII-expressing glioblastoma (ACT IV): a randomised, double-blind, international phase 3 trial. Lancet Oncol. 2017 Oct;18(10):1373-1385. doi: 10.1016/S1470-2045(17)30517-X. Epub 2017 Aug 23. PMID 28844499
- [Derived] Seliger C, Oppong FB, Lefranc F, Chinot O, Stupp R, Nabors B, Gorlia T, Weller M; EORTC Brain Tumor Group. Association of antidepressant drug use with outcome of patients with glioblastoma. Int J Cancer. 2023 Apr 1;152(7):1348-1359. doi: 10.1002/ijc.34344. Epub 2022 Nov 17. PMID 36346112